CLINICAL TRIAL: NCT01970267
Title: Randomized Trial of Laser Ablation for Highly Symptomatic Floaters
Brief Title: Clear Vision Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H13-01836
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Posterior Vitreous Detachment; Vitreous Floaters
MeSH Terms: conditions — Vitreous Detachment; vitreous floaters

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser Treated (Active Comparator): Laser will direct the laser at vitreous opacities. The power of the laser will be adjusted from 0.3-12 millijoules (mJ) with the end point being laser induced optical breakdown and the production of a small gas bubble 50% of the time. The treatment will attempt to reduced or eliminate symptomatic floaters in the visual axis. Each treatment session will be limited to 300 laser applications. Participants will be retreated based on continued symptoms for up to 5 sessions
  Interventions: Procedure: Laser Ablation of Floaters
- Not Treated (Sham Comparator)
  Interventions: Procedure: Sham Laser Treatment

INTERVENTIONS:
Procedure: Laser Ablation of Floaters
  Arms: Laser Treated
Procedure: Sham Laser Treatment — Laser will be set at 0.3 millijoules (mJ). There will be a 100% absorptive filter (black spot) of about 1cm placed centrally on the lens. All laser aiming beams will be placed within the 1cm filter. Laser will be applied at 0.3 mJ at the absorptive black spot (100% density filter) in order to create a realistic treatment therapy procedure.
  Arms: Not Treated

SUMMARY:
Vitreous floaters are tiny, cloudy, clumps of cells that appear in the otherwise clear fluid (vitreous) that fills the back 3/4 of the eye. Floaters are commonly caused by eye conditions such as posterior vitreous detachment (PVD), vitreous syneresis and asteroid hyalosis. While these symptoms are considered physiological in nature, they can be of considerable inconvenience to many patients which affect essential activities. The investigators wish to assess the safety and efficacy of floater treatment in patients with highly symptomatic floaters using an FDA approved nanosecond infrared yttrium aluminum garnet (YAG) lasers.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with symptomatic floaters lasting more than 2 months
* Willing to proceed with intervention
* Be able to provide informed consent
* Diagnosed with Posterior Vitreous Detachment
* Accept a 1% risk of complications

Exclusion Criteria:

* Less than 19 years of age
* Is a high myope (greater than -6 diopters)
* Has monocular vision
* Diagnosed with asteroid hyalosis
* Diagnosed with acute on-set of floaters (less than two months and may clear spontaneously)
* Has corneal or lenticular opacities or any media opacity which may interfere with treatment
* Has any concomitant ocular disease or pathology
* Has elevated intraocular pressure (IOP) or on IOP lowering medication
* Has floaters that are deemed to require more than five treatment sessions, where surgical intervention is the best treatment course
* Has floaters inaccessible with current lasers and lenses
* Has floaters located less than 2mm from the crystalline lens or the retina
* Found to have retinal tears or retinal detachment on initial examination or has had a history of retinal detachment repair within the last two years
* Has psychiatric problems that may recur or worsen
* Incapacity to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of the laser treatment measured by the improvement of visual acuity and floater specific Visual Function Questionnaire (VFQ). | after the last treatment session (approximately 5 days)

SECONDARY OUTCOMES:
Number of complications in the laser treated eyes compared to the non-treated eyes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B Merkur, MD, Study Chair — University of British Columbia; Mei Young, MASc, Study Director — University of British Columbia
Locations (2):
- Canada (2):
  - West Coast Retina Consultants Clinic, Vancouver, British Columbia
  - Eye Care Centre, Vancouver General Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No